CLINICAL TRIAL: NCT03693378
Title: A Prospective, Multi-center Investigational Study of IMMray™ PanCan-d Diagnostic Assay for Early Detection of Pancreatic Ductal Adenocarcinoma in High-risk Populations
Brief Title: A Study of IMMray™ PanCan-d Test for Early Detection of Pancreatic Cancer in High-risk Groups
Status: Completed | Type: Observational
Sponsor: Immunovia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PanFAM-1
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Familial Pancreatic Cancer; FAMMM - Familial Atypical Mole Malignant Melanoma Syndrome
Keywords: high-risk familial; screening program; pancreatic cancer
MeSH Terms: conditions — Pancreatic carcinoma, familial; Dysplastic Nevus Syndrome; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PanFAM-1 is a clinical study for early detection of pancreatic cancer in high-risk groups. The goals of the study are to assess the performance and diagnostic accuracy of the IMMray™ PanCan-d test compared to standard-of-care imaging.

DETAILED DESCRIPTION:
PanFAM-1 is a prospective, multi-center, investigational study, designed to assess the performance of the IMMray™ PanCan-d test in early detection of pancreatic ductal adenocarcinoma (PDAC) in high-risk populations. Specifically, the IMMray PanCan-d test uses state of the art machine learning algorithms to condense the multiple fluorescence data points generated by the test to a simple yes/no result. Thus, a highly complex statistical model uses the multi-dimensional nature of the test to generate a score, which is called a decision value. The score is compared to the established cut-off value for the test to inform the operator whether the patient sample is positive or negative for PDAC. This study will validate and evaluate the performance of the IMMray PanCan-d test in comparison to standard of care imaging approaches that are currently used in PDAC disease surveillance. Subjects in this study will be recruited from several European and North American research sites that have a PDAC surveillance program or established protocol for monitoring individuals considered to be at a high-risk for developing pancreatic cancer. Any subject that shows disease progression while on-study will be removed from the study to receive standard of care per institutional guidelines. Overall, this study poses minimal risk to subjects. The PanFAM-1 study is an adaptive study design over two approximately 18 month intervals, which are separated by an interim analysis to evaluate diagnostic accuracy of the IMMray PanCan-d test. This study is an observational period in which blood collections from eligible subjects will be evaluated using the IMMray PanCan-d test. Subjects will undergo scheduled imaging assessment and clinical evaluation consistent with the resarch sites' PDAC surveillance program. Subject data derived from the IMMray PanCan-d test during this portion of the study will be delayed from time of initial blood collection until the samples are analyzed. The analysis will compare IMMray PanCan-d test results for each subject to corresponding imaging assessments performed as part of standard of care PDAC surveillance. The study will only proceed to the interventional period if the interim analysis indicates that the diagnostic accuracy of the IMMray PanCan-d test is capable of detecting PDAC in high-risk subjects with the same or better ability as standard of care imaging. If at any time imaging assessments are considered positive for clinical disease then, regardless of IMMray PanCan-d test results, subjects will be managed according to institutional guidelines. All scheduled blood collections for purposes of this study will be halted and subjects will be removed from the study upon confirmation of PDAC.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document
2. Individuals with the following family phenotype and age:

   1. Two or more relatives with pancreatic adenocarcinomas (PDAC) on the same side of the family, where two PDAC-affected individuals are first degree related (FDR) + at least one PDAC-affected individual is a FDR of the Participant (≥50 years old OR 10 years before onset in family)
   2. Two affected FDR with PDAC (≥50 years old OR 10 years before onset of an FDR)
   3. Any of BRCA1, BRCA2, PALB2, ATM mutations confirmed pathogenic or likely pathogenic + one FDR or secondary degree related (SDR) with PDAC (≥50 years old OR 10 years before onset of an FDR and SDR)
   4. Familial atypical multiple mole-melanoma (FAMMM) with confirmed pathogenic or likely pathogenic mutation variants in: p16, CDKN2A (≥50 years old)
   5. Known mutation carrier for STK11 (Peutz Jeghers Syndrome) (≥35 years old)
   6. Lynch syndrome (HNPCC) with confirmed pathogenic or likely pathogenic variants in: MLH1, MSH2, MSH6, PMS2, or EPCAM + one FDR or SDR with PDAC (≥50 years old OR 10 years before onset of an FDR or SDR)
   7. Hereditary pancreatitis with confirmed PRSS1 pathogenic or likely pathogenic history of pancreatitis (≥40 years old)

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: High-risk patient population, enrolled in established PDAC screening programs
Sampling Method: Probability Sample
Enrollment: 1349 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Validation of IMMray™ PanCan-d test | Approximately 18 months upon collection of approximately 2,000 subjects, or disease progression, whichever comes first
  Demonstrate that the IMMray PanCan-d test is equal or better than the reference standard imaging procedures for early detection of PDAC in asymptomatic high risk individuals

SECONDARY OUTCOMES:
Evaluation of the IMMray™ PanCan-d test performance | Approximately 18 months upon collection of approximately 2,000 subjects, or disease progression, whichever comes first
  Point Estimates and 95% confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Ehrnström, Study Director — Immunovia, Inc.
Locations (21):
- United States (13):
  - Stanford Gastroenterology and Hepatology, Stanford, California
  - Yale University, New Haven, Connecticut
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - New York University Hospital, New York, New York
  - Columbia University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- The Research Institute of the McGill University Health Centre, Montreal, Canada
- Spain (2):
  - University Hospital Ramon y Cajal, Madrid
  - University Hospital Santiago De Compostela, Santiago de Compostela
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm
  - Umeå University Hospital, Umeå
- University Collage London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mellby LD, Nyberg AP, Johansen JS, Wingren C, Nordestgaard BG, Bojesen SE, Mitchell BL, Sheppard BC, Sears RC, Borrebaeck CAK. Serum Biomarker Signature-Based Liquid Biopsy for Diagnosis of Early-Stage Pancreatic Cancer. J Clin Oncol. 2018 Oct 1;36(28):2887-2894. doi: 10.1200/JCO.2017.77.6658. Epub 2018 Aug 14. PMID 30106639
- [Derived] Brand RE, Persson J, Bratlie SO, Chung DC, Katona BW, Carrato A, Castillo M, Earl J, Kokkola A, Lucas AL, Moser AJ, DeCicco C, Mellby LD, King TC. Detection of Early-Stage Pancreatic Ductal Adenocarcinoma From Blood Samples: Results of a Multiplex Biomarker Signature Validation Study. Clin Transl Gastroenterol. 2022 Feb 14;13(3):e00468. doi: 10.14309/ctg.0000000000000468. PMID 35166713
- [Derived] Abstracts of Papers Submitted to the 52nd Meeting of the American Pancreatic Association, November 3-6, 2021, Miami Beach, Florida. Pancreas. 2021 Aug 1;50(7):1044-1115. doi: 10.1097/MPA.0000000000001904. No abstract available. PMID 34643612